CLINICAL TRIAL: NCT04037527
Title: Phase I Trial Study of Gemcitabine and Docetaxel With Radiation in Adult Patients With High Grade and Greater Than 5 cm Soft Tissue Sarcoma of the Extremities
Brief Title: Gemcitabine and Docetaxel With Radiation in Adults With Soft Tissue Sarcoma of the Extremities
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due DLTs
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061621; P30CA012197 (NIH); CCCWFU 71117 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Soft Tissue Sarcoma
Keywords: Grade II sarcoma; Grade III sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Docetaxel; Radiation; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Chemotherapy Plus Radiation Therapy (Experimental): Up to 6 cycles (once a week) of chemotherapy with a 3+3 dose escalating plan (from 100 mg to 300 mg for Gemcitabine; 10 mg to 25 mg for Docetaxel) along with radiation (five days a week) for up to 6 weeks.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Radiation: Radiation; Procedure: Surgical Resection; Other: Blood draws

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be administered on day 1 of each one-week cycle for 6 cycles concurrently with radiation to the extremity on a 3+3 escalating dose (100 mg/m² to 300 mg/m²)
Drug: Docetaxel — Docetaxel will be administered on day 1 of each one-week cycle for 6 cycles concurrently with radiation to the extremity (10 mg/m² to 25 mg/m²).
  Other Names: Taxotere
Radiation: Radiation — Radiation is to be done with standard preop dose of 50 Gy but at lower doses per fraction. Thus 50.4 Gy in 28 FX. Radiation will be given for 5 days (Monday - Friday) every week for approx. 6 weeks.
Procedure: Surgical Resection — Upon completing neoadjuvant chemotherapy plus radiation therapy, surgical resection will occur.
Other: Blood draws — Before treatment, blood (about 2 tubes of 10 mls each) to better understand some aspects of participants' immune system before chemotherapy.

SUMMARY:
The purpose of this Phase 1 research study is to obtain data or information on the safety and effectiveness of the combination of gemcitabine, docetaxel with radiation.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the maximum tolerated doses Gemcitabine and Taxotere when given weekly with concurrent radiation in the neoadjuvant setting for patients with soft tissue sarcoma of the extremities.

Secondary Objective:

• To evaluate immunological changes induced by gemcitabine and docetaxel with radiation in patient with high risk-soft tissue sarcomas in blood. This would include T cell subsets, NK, and dendritic cells and tumor macrophages all of which make up the tumor microenvironment.

Long term follow-up will occur every 3-4 months for 24 months in person or video consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed Grade II or III soft tissue sarcoma that is considered to be resectable and are candidates for pre-op radiation.
* Age greater than or equal to 18 years. No children will be enrolled on this protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or double-barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients taking concurrent hormonal therapy, biologic or other chemotherapy are excluded except women on hormonal contraceptives.
* Patients taking an investigational agent are excluded.
* Pregnant and nursing women are excluded.
* Patients who require amputation for local control.
* Patients who underwent unplanned excision or other previous surgery involving the affected extremity.
* Patients with sarcoma subtypes for which established chemotherapeutic regimens exist.
* History of radiation to the limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose Chemotherapy and Radiation | Up to 8 weeks
  Maximum tolerated dose of Gemcitabine and Taxotere and radiation will be completed by monitoring toxicities and using the 3+3 dose escalation plan.
Number of Toxicity Incidences | 8 weeks post-surgery
  Complication/side effects from the chemotherapy combination of gemcitabine and taxotere concurrent with radiation will be assessed by toxicity counts/rates presented descriptively by toxicity, severity, and dose level using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Number of Immunological Changes in Blood | 8 weeks post-surgery
  The effects of the treatment on the immune system will be analyzed using paired t-test or the non-parametric counterpart. Correlations between immune cells and immune factor levels will be assessed using Spearman correlation coefficient. All tests will be two-sided with a significance level of 0.05, and no adjustment for multiple comparisons will be made due to the exploratory nature of these studies.

CONTACTS AND LOCATIONS:
Overall Officials: Shailaja Raj, MRCP, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04037527/ICF_000.pdf